CLINICAL TRIAL: NCT05083702
Title: Ultrasound Versus Fluoroscopic Guided Superior Hypogastric Plexus Block in Cancer Bladder: A Randomized Controlled Trial
Brief Title: Ultrasound Versus Fluoroscopy Guided Superior Hypogastric Plexus Block in Cancer Bladder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AP2103-30101R
Record Dates: First submitted 2021-06-10; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Pain, Chronic
Keywords: fluroscopy and ultrasound SHPB in cancer bladder
MeSH Terms: conditions — Chronic Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluoroscopy-guided superior hypogastric plexus block transdiscal approach (Active Comparator): fluroscopy guided superior hypogastric plexus block transdiscal approach for chronic pain treatment in cancer bladder VAS score and morphine consumption are measured before and after 1 day , 1 month , 3 monthes
  Interventions: Procedure: Fluoroscopy-guided superior hypogastric plexus block transdiscal approach
- ultrasound-guided superior hypogastric plexus block (Active Comparator): ultrasound guided superior hypogastric plexus block in treatment of chronic pain in cancer badder VAS score and morphine consumption are measured before and after 1 day , 1 month , 3 monthes
  Interventions: Procedure: ultrasound-guided superior hypogastric plexus block

INTERVENTIONS:
Procedure: Fluoroscopy-guided superior hypogastric plexus block transdiscal approach — Patient lies prone, L5-S1 interspace identified under fluoroscopy, the skin is prepared and sterile drapes are placed after local anesthetic infiltration of the skin the subcutaneous tissue with 2% lidocaine a 20 guage, 15 cm needle with short bevel is inserted at the center of L5- S1 interlaminar space under anteroposterior fluoroscopic vision. The needle is then advanced toward the intervertebral disc. After confirmation, the needle is advanced through the intervertebral disc until it exists at its anterior surface confirmed by administration of 4 ml of soluble contrast media in both lateral and anteroposterior fluoroscopic view. Neurolysis is performed with 8 ml 8 % phenol solution. After neurolysis, 0.5 ml of saline is given to avoid the deposition of phenol within the intervertebral disc material. While withdrawing, the needle cephazoline 50 mg in 1 ml is injected into the disc.
  Other Names: fluroscopy
  Arms: Fluoroscopy-guided superior hypogastric plexus block transdiscal approach
Procedure: ultrasound-guided superior hypogastric plexus block — Patients are placed in the supine position and after sterilization, the low-frequency curved probe is used in the longitudinal axis to visualize the aortic bifurcation and is identified using a longitudinal Ultra-Sound (Phillips Healthcare, Andover, Massachusetts, US). Next, the probe is placed deeply transverse till aorta end and bifurcation seen of iliac vessels once seen we enter out of plane and inject.as it lies in front the vertebral body of the L5 vertebra. Local infiltration with 1% lidocaine is obtained at port of entry 1-1.5 inches below the umbilicus. A 15-cm, 22-G Chiba needle is inserted (out-of-plane) and advanced by avoiding vascular structures until contact with the L5-body. The needle will be withdrawan the 1-2 mm and inject 8 ml 8% phenol in saline. Finally, 0.5 ml of lidocaine is injected during Chiba needle removal
  Other Names: ultrasound
  Arms: ultrasound-guided superior hypogastric plexus block

SUMMARY:
Pelvic cancer pain is a chronic condition related to the involvement of viscera, pelvic muscular structures or neural structures by tumor. The superior hypogastric plexus block is a sympathetic block used to treat pelvic visceral pain that is unresponsive to oral or parenteral opioids different approaches for superior hypogastric block as transdiscal approach, classic approach, Posteromedial approach, CT guided approach and ultrasound anterior approach The ultrasound-guided superior hypogastric plexus neurolysis technique (anterior approach) is simple to perform. We believe this block can be useful in cancer patients who are having difficulty in lying prone, because it is a procedure performed in the supine position and it is less time-consuming. It also avoids the radiation exposure involved with a computed tomography-guided and fluoroscopy posterior approach.

DETAILED DESCRIPTION:
Aim of the study:

To compare Fluoroscopic guided transdiscal superior hypogastric block and Ultrasound guided superior hypogastric block regarding their efficacy to control pelvic pain and

Statistical analysis:

Data will be described as mean ±SD or as frequencies (number of cases) and percentages when appropriate. Comparison of numerical variables between two study groups will be carried out using parametric and non-parametric t- tests for independent samples. Within group comparison of numerical variables was carried out using repeated measures ANOVA. P values of less than 0.05 will be statistically significant. All statistical calculations are performed using statistical package for the social sciences (SPSS, version 23 for Microsoft Windows; SPSS Inc., Chicago, Illinois, USA)

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years.
* Patients with advanced stage cancer bladder.
* Patient with severe pain (VAS) 7 or more .
* Patients don't receive any strong opioids for pain at least 2 weeks

Exclusion Criteria:

* Patient refusal.
* Local infection at the puncture site.
* Coagulopathy.
* Cognitive disorders.
* Unstable cardiovascular disease.
* History of psychiatric disorders.
* History of drug abuse.
* Patients allergic to medication used.
* Patients with any contraindications to drugs and dye used.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score | Three months after the procedure
  Pain Intensity measured by Visual analogue scale score16 (A 100 mm horizontal line version is used with 2 ends left end means no pain and right end means the worst pain.
  VAS will be recorded before and after the procedure, at the first day, after 1 month and after 3 months.

SECONDARY OUTCOMES:
The amount of daily morphine consumption | Three months after the procedure
  Daily morphine or other drugs consumption according to WHO ladder after the procedure.
  This will be recorded before and after the procedure, at the first day, after 1 month and after 3 months.
Patient functional capacity | Three months after the procedure
  Patient functional capacity (is evaluated using Eastern cooperative oncology group "ECOG" scoring (0=fully active, 1= able to perform light effort, 2= in bed <50% of the day 3=in bed >50% of the day, 4=bed ridden).
  This will be recorded before and after the procedure, at the first day, after 1 month and after 3 months.
Quality of life | Three months after the procedure
  Patient quality of life SF-36 19 (consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  This will be recorded before and after the procedure, at the first day, after 1 month and after 3 months.
Complications | Three months after the procedure
  Any complications will be detected: back pain, bleeding, infection, L5 root injury with paresthesia or motor weakness, and visceral or vascular injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Mostafa, Study Director — National Cancer Institute (NCI)
Locations (1):
- National cancer institute, Cairo, Egypt